CLINICAL TRIAL: NCT00788476
Title: Needs Assessment Survey in Childhood Cancer Survivors and Their Parents
Brief Title: Childhood Cancer Survivor Survey
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0490
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2013-10

CONDITIONS: Cancer
Keywords: Needs Assessment Survey; Childhood Cancer Survivors; Parents; Primary Caregiver; Survey
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Childhood Cancer Survivors
  Interventions: Other: Survey
- Primary Caregivers
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey packets to adult (>18 years old) childhood cancer survivors who return to MDACC for follow-up appointments within the next 12-months and conduct a mailed survey with the remaining participants and their "primary caregivers" i.e. guardians of survivors who are currently under age 18.
  Other Names: Questionnaire

SUMMARY:
Objectives:

1. To explore current lifestyle practices, health status, and quality of life among childhood cancer survivors and parent/guardians who are identified as "primary caregivers."
2. To explore childhood cancer survivors' and "primary caregivers'" awareness of future health risks.
3. To explore interest in various lifestyle interventions and delivery channels among childhood cancer survivors and their "primary caregivers."
4. To explore factors which may serve as mediators or moderators of future lifestyle interventions that target childhood cancer survivors and their "primary caregivers," e.g., strength of the caregiver-child bond, geographic distance from one another, and level of education.

DETAILED DESCRIPTION:
A mailed survey will be conducted that will assess the health behaviors (diet, exercise, and tobacco-use) of childhood cancer survivors, and the behaviors of identified "primary caregivers" (see definition under inclusion criteria). In addition, these surveys will assess awareness of longterm health risks, quality of life (QOL), strength of the child-caregiver bond, body image, body weight status, functional status, barriers to lifestyle change, and interest in various lifestyle interventions and potential channels for delivery. Mailed surveys (with telephone follow-up) will be sent to MDACC childhood cancer survivors diagnosed from 1998 - 2007 who are survivors of central nervous system (CNS) tumors, sarcomas, lymphoma or leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for childhood cancer survivors: 1) diagnosed between 1992-2007 with central nervous system tumors, sarcomas, leukemia, or lymphoma; 2) off active treatment for at least six-months, and alive with no evidence of progressive disease; 3) currently between age 8 (i.e., at an age at which they could be reasonably expected to complete a survey and where validated instruments exist) and 34 (cutpoint based on the possibility that individuals were almost 18 in 1992 and decade has since passed); and 4) able to speak or read English.
2. Inclusion criteria for parents/guardians: 1) parents/guardians of childhood cancer survivors diagnosed from 1992-2007 with central nervous system tumors, sarcomas, leukemia, or lymphoma who completed active treatment at least six-months ago and who currently are alive with no evidence of disease; 2) parents/guardians of a survivor who is currently 2-34 years of age; 3) self-identified as the current "primary caregiver" of the survivor if the survivor is age 2-17 OR identified by the survivor as the "primary caregiver" if the survivor is age 18-34; and 4) able to speak or read English.

Exclusion Criteria:

1. Exclusion criteria for childhood cancer survivors: 1) diagnosed with cancers other than central nervous system tumors, sarcomas, leukemia, or lymphoma; 2) diagnosed with cancer either prior to 1992 or after 2007; 3) currently on treatment; 4) currently diagnosed with progressive cancer; 5) deceased; 6) under age 8 or over age 34; or 7) non-English speaking or reading.
2. Exclusion criteria for parent/guardians: 1) parent/guardians of childhood cancer survivors who were diagnosed with cancer before 1992 or after 2007 OR with cancers other than CNS tumors, sarcomas, leukemia, or lymphoma OR whose children are currently on treatment, have progressive cancer or are deceased OR whose children are currently <2 or >34 years old; 2) non-English speaking/reading; or 3) do not self-identify as being the current "primary caregiver" of childhood cancer survivors ages 2-17 or are not identified as being the primary caregiver of childhood cancer survivors who are age 18+.

Ages: 8 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Childhood cancer survivors between ages of 8 and 28 years of age and their primary caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2008-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Patient Response Rate to Survey | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Joann L. Ater, MD, BA, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org